CLINICAL TRIAL: NCT05416827
Title: Evaluation of Intraoperative Slow-release Dexamethasone Implant Used During Vitrectomy for Epiretinal Membrane
Brief Title: Evaluation of Intraoperative Slow-release Dexamethasone Implant for Epiretinal Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PKUPHophthal
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Epiretinal Membrane
Keywords: Epiretinal Membrane; Ozurdex; PPV
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPV group (Active Comparator): Epiretinal membrane eyes underwent PPV
  Interventions: Procedure: slow-release dexamethasone implant
- PPV+implant Group (Experimental): Epiretinal membrane eyes underwent PPV combined with Ozurdex implant
  Interventions: Procedure: slow-release dexamethasone implant

INTERVENTIONS:
Procedure: slow-release dexamethasone implant — Epiretinal membrane eyes underwent PPV combined with Ozurdex implant

SUMMARY:
Epiretinal membrane (ERM) is a commonly encountered vitreoretinal interface anomaly with a prevalence of approximately 10% in the adult population. It is often treated with pars plana vitrectomy (PPV) and membrane peeling when symptomatic. PPV is generally successful at improving visual acuity (VA) and/or metamorphopsia. At times, however, visual recovery can be hindered by macular edema in the post-vitrectomy period. Ozurdex can accelerate the resorption of intraretinal edema and hasten the improvement in the visual acuity. It has been shown to facilitate fluid absorption by both stimulating endogenous adenosine signaling in Muller cells and by down regulating vascular endothelial growth factor production. So, this study aim to investigate the efficacy of Ozurdex implant after PPV in epiretinal membrane eyes.

DETAILED DESCRIPTION:
Small gauge pars plana vitrectomy (PPV) with membrane peeling is used to successfully treat macular epiretinal membranes (ERMs) with a postoperative improvement of visual acuity in the majority of cases. Traditionally, the treatment of ERMs has been performed purely by peeling the membrane mechanically and then waiting for the intraretinal edema to resolve spontaneously. In the last few years, some publications raised the possibility that triamcinolone acetonide (TA),given as an intravitreal injection at the end of surgery, can accelerate the resorption of intraretinal edema and hasten the improvement in the visual acuity. It has been shown to facilitate fluid absorption by both stimulating endogenous adenosine signaling in Muller cells and by down regulating vascular endothelial growth factor production. Dexamethasone is a potent synthetic member of the glucocorticoid class of steroid drugs that has anti-inflammatory and immunosuppressant activity 30 times that of cortisol and 6 times that of triamcinolone. As the postoperative cystoid macular edema usually peaks 4 to 6 weeks after surgery the difference in the half life can be significant and explained the results in past publications. While the use of intravitreal TA as an adjuvant to PPV with membrane peel showed conflicting results. Only few publications demonstrated the effectiveness of Ozurdex in the treatment of macular edema in a vitrectomized eye, after ERM removal.So, this study aim to investigate the efficacy of Ozurdex implant after PPV in epiretinal membrane eyes.

ELIGIBILITY:
Inclusion Criteria:

* patients with a visually significant (BCVA<20/50) idiopathic epiretinal membrane.
* ocular axial length less than 27.00 mm (optical biometry) associated with cataracts.

Exclusion Criteria:

* concomitant or previous macular diseases (diabetic macular edema, retinal vein occlusion and agerelated macular degeneration).
* secondary epiretinal membrane, other visually significant macular pathology and prior intravitreal triamcinolone acetonide injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
CMT | from preoperation to 3 months follow-up
  central macular thickness
IOP | from preoperation to 3 months follow-up
  intraocular pressure
BCVA | from preoperation to 3 months follow-up
  best-corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Jinfeng Qu, MD, Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reilly G, Melamud A, Lipscomb P, Toussaint B. SURGICAL OUTCOMES IN PATIENTS WITH MACULAR PUCKER AND GOOD PREOPERATIVE VISUAL ACUITY AFTER VITRECTOMY WITH MEMBRANE PEELING. Retina. 2015 Sep;35(9):1817-21. doi: 10.1097/IAE.0000000000000558. PMID 25923959
- [Background] Mao J, Xu Z, Lao J, Chen Y, Xu X, Wu S, Zheng Z, Liu B, Shen L. Assessment of macular microvasculature features before and after vitrectomy in the idiopathic macular epiretinal membrane using a grading system: An optical coherence tomography angiography study. Acta Ophthalmol. 2021 Nov;99(7):e1168-e1175. doi: 10.1111/aos.14753. Epub 2021 Jan 10. PMID 33423352
- [Background] Yang HS, Kim JT, Joe SG, Lee JY, Yoon YH. Postoperative restoration of foveal inner retinal configuration in patients with epiretinal membrane and abnormally thick inner retina. Retina. 2015 Jan;35(1):111-9. doi: 10.1097/IAE.0000000000000276. PMID 25102192
- [Background] Beer PM, Bakri SJ, Singh RJ, Liu W, Peters GB 3rd, Miller M. Intraocular concentration and pharmacokinetics of triamcinolone acetonide after a single intravitreal injection. Ophthalmology. 2003 Apr;110(4):681-6. doi: 10.1016/S0161-6420(02)01969-3. PMID 12689886
- [Background] Chin HS, Park TS, Moon YS, Oh JH. Difference in clearance of intravitreal triamcinolone acetonide between vitrectomized and nonvitrectomized eyes. Retina. 2005 Jul-Aug;25(5):556-60. doi: 10.1097/00006982-200507000-00002. PMID 16077349
- [Background] Medeiros MD, Alkabes M, Navarro R, Garcia-Arumi J, Mateo C, Corcostegui B. Dexamethasone intravitreal implant in vitrectomized versus nonvitrectomized eyes for treatment of patients with persistent diabetic macular edema. J Ocul Pharmacol Ther. 2014 Nov;30(9):709-16. doi: 10.1089/jop.2014.0010. Epub 2014 Sep 26. PMID 25259834
- [Background] Boyer DS, Faber D, Gupta S, Patel SS, Tabandeh H, Li XY, Liu CC, Lou J, Whitcup SM; Ozurdex CHAMPLAIN Study Group. Dexamethasone intravitreal implant for treatment of diabetic macular edema in vitrectomized patients. Retina. 2011 May;31(5):915-23. doi: 10.1097/IAE.0b013e318206d18c. PMID 21487341
- [Derived] Li S, Zeng Q, Zhu L, Liu W, Li Y, Li J, Li X, Zhao M, Qu J. Intraoperative slow-release dexamethasone intravitreal implant (Ozurdex) in epiretinal membrane peeling surgery: a prospective randomized controlled trial. Front Pharmacol. 2023 Sep 1;14:1219861. doi: 10.3389/fphar.2023.1219861. eCollection 2023. PMID 37727387